CLINICAL TRIAL: NCT04489238
Title: Young Onset Gastrointestinal Cancer Prospective Registry
Brief Title: Collection of Information to Better Understand Young Onset Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-315
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma
Keywords: young onset colorectal cancer; colorectal registry; 20-315; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young onset Colorectal Cancer Participants: (Stool collection on newly diagnosed patients in this cohort) Participants will include patients under the age of 50 who are diagnosed with colorectal adenocarcinoma.
  Interventions: Other: Risk Factor Questionnaire
- Average onset Colorectal Cancer Participants: (Stool collection cohort only) 166 colorectal cancer patients 50 year-old or older will serve as controls.
  Stool collection cohort only.
  Interventions: Other: Risk Factor Questionnaire

INTERVENTIONS:
Other: Risk Factor Questionnaire — Participants, both cases and controls, will complete the CYOC risk factor questionnaire, preferably at the time of first visit
  Other Names: CYOC Risk Factor Questionnaire

SUMMARY:
The purpose of this registry study is to create a database-a collection of information-for better understanding young onset colorectal cancer. Colorectal cancer patients are considered to have young onset colorectal cancer if they are diagnosed with their cancer before the age of 50. Researchers will use the information from this database to learn more about how young onset colorectal cancer may be similar to or different from colorectal cancer that is diagnosed later in life. Researchers will also use information from the database for current and future research on young onset colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria for database and questionnaire (YOGI)

* Histological or cytological diagnosis of gastrointestinal cancer
* 18 - 49 years old at time of consent
* No Known hereditary CRC or other cancer predisposition syndrome (stool collection cohort only)
* No history of inflammatory bowel disease (stool collection cohort only)
* No prior diagnosis of gastrointestinal cancer (stool collection cohort only)

Participant Inclusion Criteria for database and questionnaire (Controls)

* Histological or cytological diagnosis of colorectal adenocarcinoma
* No previous treatment for CRC (including surgery, chemotherapy, immunotherapy or radiation)
* Age 50 or older at time of consent
* No Known hereditary CRC or other cancer predisposition syndrome
* No history of inflammatory bowel disease
* No prior diagnosis of CRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified through the Center for Young Onset Gastrointestinal Cancer, a member of the patient's treatment team, the principal investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC). All study participants will be recruited from patients under the care of consenting professionals. If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Probability Sample
Enrollment: 1366 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Establish a prospective database of patients with Young Onset Colorectal Cancer | 1 year
  from diagnosis through survivorship

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - MSK at Ralph Lauren, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org